CLINICAL TRIAL: NCT04208724
Title: Implementation Studio, an Innovative, Structured Approach to Facilitate Rural Community-Based Organizations' Adaptation and Implementation of Evidence-Based Interventions
Brief Title: Support Program for Adoption of Cancer Screening Interventions at a Rural Community-Based Organization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RG1006143; NCI-2019-08033 (Registry Identifier: NCI / CTRP); 10307 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-12-10; First posted 2019-12-23 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Breast Carcinoma; Cervical Carcinoma; Colorectal Carcinoma; Malignant Solid Neoplasm
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Colorectal Neoplasms | interventions — Resistance Training; Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training program (Experimental): Community-based organizations participate in the support program, consisting of 2 half-day training workshops over 2 weeks, and 30-minute bi-weekly consultations in order to adapt and implement the cancer screening intervention for community members.
  Interventions: Other: Training; Other: Cancer Screening intervention; Other: Survey Administration

INTERVENTIONS:
Other: Training — Participate in the training program
  Other Names: Training Programs
Other: Cancer Screening intervention — Receive cancer screening intervention
  Other Names: cancer screening
Other: Survey Administration — Ancillary studies

SUMMARY:
This pilot trial study uses a structural support program for adoption of cancer screening interventions at a rural community-based organization. Rural communities face unique barriers in implementation of evidence-based interventions due to a lack of infrastructure, community capacity, and expertise as academic and research centers are often clustered in urban areas. The support program may help a rural community-based organization select, adapt, and implement cancer prevention and control evidence-based interventions.

DETAILED DESCRIPTION:
OUTLINE:

Community-based organizations participate in the support program, consisting of 2 half-day training workshops over 2 weeks, and 30-minute bi-weekly consultations in order to adapt and implement the cancer screening intervention for community members.

After completion of study, participants are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Objective II COMMUNITY-BASED ORGANIZATION: Located in the Yakima Valley of Washington State
* Objective II COMMUNITY-BASED ORGANIZATION: Serve community members who are 18 and older
* Objective II COMMUNITY-BASED ORGANIZATION: Willing to commit to the 6-month program
* Objective II PARTICIPANTS: Receiving services from the recruited community-based organization
* Objective III PARTICIPANTS: Not up-to-date for breast, cervical, and colorectal cancer screening according to current U.S. Preventive Services Tasks Force (USPSTF) guidelines. The current USPSTF recommendations for breast, cervical, and colorectal cancer are:

  * Breast Cancer Screening: Women ages 50-74 should be screened for breast cancer with mammography every 2 years.
  * Cervical Cancer Screening: Women ages 21-29 should be screened for cervical cancer every 3 years with cervical cancer cytology alone. For women ages 30-65, the USPSTF recommends screening every 3 years with cervical cytology alone, every 5 years or every 5 years with high risk human papillomavirus (hrHPV) testing in combination of cytology.
  * Colorectal Cancer Screening: Individuals ages 50-75 should be screened for colorectal cancer with guaiac-based fecal occult blood tests (gFOBT) or fecal immunochemical test (FIT) once a year, or colonoscopy every 10 years (USPSTF approves additional screening tests, but these are the most commonly used).
* Objective III PARTICIPANTS: If the community-based organization selects breast cancer screening, we will recruit women ages 50-74.
* Objective III PARTICIPANTS: If the community-based organization selects cervical cancer screening, we will recruit women ages 21-65.
* Objective III PARTICIPANTS: If the community-based organization selects colorectal cancer screening, we will recruit women and men ages 50-75.
* Objective III PARTICIPANTS: Average risk for breast, cervical, or colorectal cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Develop the structural program | 3 months
  Development of the structural training program and accompanying tools
Implementation Monitoring | 4 months
  Implementation of the evidence-based intervention by the community-based organization including 1) dosage (how many interventions were delivered to the participants), 2) types (for which cancer), 3) length of exposure (for how long), and 4) who is involved in the implementation (by whom).
Intention to get screened for cancer (type of cancer will be determined by the community-based organization) pre- and post-intervention | Up to 3 months
  Difference in the proportion of intention to get screened for cancer pre- and post-intervention using chi-square analyses

CONTACTS AND LOCATIONS:
Overall Officials: Linda Ko, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ko LK, Vu T, Bishop S, Leeman J, Escoffery C, Winer RL, Duran MC, Masud M, Rait Y. Implementation studio: implementation support program to build the capacity of rural community health educators serving immigrant communities to implement evidence-based cancer prevention and control interventions. Cancer Causes Control. 2023 Dec;34(Suppl 1):75-88. doi: 10.1007/s10552-023-01743-6. Epub 2023 Jul 13. PMID 37442868

DOCUMENTS (1):
  • Informed Consent Form (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT04208724/ICF_000.pdf